CLINICAL TRIAL: NCT03411317
Title: Aortic Stenosis: Determinants of Progression, Severity and Left Ventricular Remodeling (AS-PROGRESSION)
Brief Title: Aortic Stenosis: Determinants of Progression, Severity and Left Ventricular Remodeling
Acronym: AS-PROGRESSION
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Rouen (Other)
Responsible Party: Sponsor
Other Study IDs: 2017/081/HP
Record Dates: First submitted 2017-08-21; First posted 2018-01-26 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Aortic Valve Stenosis
Keywords: Aortic stenosis; progression; Left ventricular remodeling
MeSH Terms: conditions — Aortic Valve Stenosis; Disease Progression; Ventricular Remodeling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Aortic stenosis (AS) is the most frequent valvulopathy in Western countries. The prevalence of AS is constantly increasing due to the aging of the population. Although significant progress has been made in understanding the pathophysiological mechanisms underlying the onset and progression of AS, there is no medical treatment to slow or prevent its progression. The only treatment available is Aortic Valve Replacement (AVR) performed by surgery or by catheterization (TAVI).

AS is associated with an increase of post-load which leads the left ventricular myocardium to hypertrophy. Associated with hypertrophy, myocardial fibrosis will gradually develop. Despite interesting data, many unknowns persist and remain to be identified.

The aim of the study is to evaluate prospectively the progression and impact of AS in 500 patients using clinical, biological, echocardiographic and MRI parameters performed annually.

ELIGIBILITY:
Inclusion Criteria:

* Aortic stenosis (peak aortic valve velocity (Vmax) ≥2.5m/s )

Exclusion Criteria:

* rheumatismal or congenital aortic stenosis
* aortic insufficiency (grade >= 2/4)
* Associated valvulopathy (grade >= 2/4)
* Angina, syncope, dyspnea NYHA 3-4
* Heart failure antecedent
* Myocardial infarction antecedent
* Severe renal failure
* indication of Aortic Valve Replacement (Surgery or TAVI)
* Cardiac surgery (Aorta abdominal) antecedent
* Complex congenital cardiopathy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with at least moderate aortic stenosis and in whom an intervention is not programmed or indicated
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2017-12-11 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Composite primary endpoint: haemodynamic and anatomical progression of Aortic Stenosis | Year 1
  CT scan and MRI
Composite primary endpoint: haemodynamic and anatomical progression of Aortic Stenosis | Year 2
  CT scan and MRI
Composite primary endpoint: haemodynamic and anatomical progression of Aortic Stenosis | Year 3
  CT scan and MRI
Composite primary endpoint: haemodynamic and anatomical progression of Aortic Stenosis | Year 4
  CT scan and MRI

SECONDARY OUTCOMES:
Determinants of left ventricular remodeling | Year 1
  MRI and echocardiography
Determinants of left ventricular remodeling | Year 2
  MRI and echocardiography
Determinants of left ventricular remodeling | Year 3
  MRI and echocardiography
Determinants of left ventricular remodeling | Year 4
  MRI and echocardiography
Progression of left ventricular remodeling | Year 1
  MRI and echocardiography
Progression of left ventricular remodeling | Year 2
  MRI and echocardiography
Progression of left ventricular remodeling | Year 3
  MRI and echocardiography
Progression of left ventricular remodeling | Year 4
  MRI and echocardiography
Prognostic value of ventricular mass, type of ventricular remodeling and fibrosis in Aortic Stenosis | Year 1
  Occurrence of clinical events, MRI, CT scan and echocardiography
Prognostic value of ventricular mass, type of ventricular remodeling and fibrosis in Aortic Stenosis | Year 2
  Occurrence of clinical events, MRI, CT scan and echocardiography
Prognostic value of ventricular mass, type of ventricular remodeling and fibrosis in Aortic Stenosis | Year 3
  Occurrence of clinical events, MRI, CT scan and echocardiography
Prognostic value of ventricular mass, type of ventricular remodeling and fibrosis in Aortic Stenosis | Year 4
  Occurrence of clinical events, MRI, CT scan and echocardiography

CONTACTS AND LOCATIONS:
Overall Officials: Helene Eltchaninoff, Pr, Principal Investigator — University Hospital, Rouen
Locations (1):
- UH Rouen, Rouen, France